CLINICAL TRIAL: NCT02779413
Title: A Multi-centre, Prospective, Open-label, Single-arm, Non-interventional, Regulatory Post Marketing Surveillance (rPMS) Study of Tresiba® FlexTouch® (Insulin Degludec) to Evaluate Safety and Effectiveness in Patients of All Age Groups Excluding Less Than 12 Months Old Infants With Diabetes Mellitus in Routine Clinical Practice in Korea
Brief Title: A Study to Evaluate Safety and Effectiveness in Patients of All Age Groups Excluding Less Than 12 Months Old Infants With Diabetes Mellitus in Routine Clinical Practice in Korea
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-4110; U1111-1176-2287 (Other: WHO)
Record Dates: First submitted 2016-05-13; First posted 2016-05-20 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin degludec
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Patients will be treated with commercially available Tresiba® FlexTouch® according to routine clinical practice at the discretion of the treating physician.

SUMMARY:
This study is conducted in Asia. The aim of the study is to evaluate safety and effectiveness in patients of all age groups excluding less than 12 month old infants with diabetes mellitus in routine clinical practice in Korea.

ELIGIBILITY:
Inclusion Criteria: - Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol) - The decision to initiate treatment with commercially available Tresiba® FlexTouch® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study - Male or Female, Age at least 12 months, at the time of signing informed consent with type 1 or type 2 diabetes mellitus and who is scheduled to start treatment with Tresiba® FlexTouch® based on the clinical judgment of their treating physician as specified in the Korean-Prescribing Information (KPI) Exclusion Criteria: - Previous participation in this study. Participation is defined as having given informed consent in this study - Patients who are or have previously treated with Tresiba® FlexTouch® - Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation. However, paediatric patients can be enrolled when the patient's primary caregiver (e.g. parents) or legally acceptable representatives (LAR) are capable of giving study specific signed informed consent. Any chronic disorder or severe disease which in the opinion of the investigator might jeopardise patient's safety or compliance with the protocol - Female who is pregnant, breast-feeding or intends to become pregnant and is of child-baring potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice)

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus requiring insulin therapy for whom it has been decided to start with Tresiba® FlexTouch® based on the clinical judgment by their treating physician will be enrolled during enrolment period
Sampling Method: Non-Probability Sample
Enrollment: 3303 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AE) | Week 13± 2 weeks
Number of Adverse Events (AE) | week 26± 2 weeks

SECONDARY OUTCOMES:
Insulin dose changes | Week 0, Week 26
Change in HbA1c | Week 0, week 13, week 26
Percentage of patients achieving the target of HbA1c below 7.0% | At week 13
Percentage of patients achieving the target of HbA1c below 7.0% | At week 26
Change in fasting plasma glucose (FPG) | Week 0, week 13, week 26
Changes in postprandial plasma glucose (PPG) | Week 0, week 13, week 26
Number of Adverse reactions (AR) | Week 13± 2 weeks
Number of Adverse reactions (AR) | week 26± 2 weeks
Number of Serious AE | Week 13± 2 weeks
Number of Serious AE | week 26± 2 weeks
Number of Serious AR | Week 13± 2 weeks
Number of Serious AR | week 26± 2 weeks
Number of Unexpected AR | Week 13± 2 weeks
Number of Unexpected AR | week 26± 2 weeks
Number of Severe hypoglycaemia (PG (plasma glucose) below 56 mg/dl) | Week 13± 2 weeks
Number of Severe hypoglycaemia (PG (plasma glucose) below 56 mg/dl) | week 26± 2 weeks
Number of Blood glucose (BG) confirmed hypoglycaemia (PG below 56 mg/dl) | Week 13± 2 weeks
Number of Blood glucose (BG) confirmed hypoglycaemia (PG below 56 mg/dl) | week 26± 2 weeks
Weight gain | week 13 ± 2 weeks
Weight gain | week 26± 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (18):
- South Korea (18):
  - Novo Nordisk Investigational Site, Bucheon-si
  - Novo Nordisk Investigational Site, Busan
  - Novo Nordisk Investigational Site, Chungcheongnam-do
  - Novo Nordisk Investigational Site, Daegu
  - Novo Nordisk Investigational Site, Daejeon
  - Novo Nordisk Investigational Site, Gangwon-do
  - Novo Nordisk Investigational Site, Gyeonggi-do
  - Novo Nordisk Investigational Site, Gyeongsangbuk-do
  - Novo Nordisk Investigational Site, Gyeongsangnam-do
  - Novo Nordisk Investigational Site, Incheon
  - Novo Nordisk Investigational Site, Jeonju
  - Novo Nordisk Investigational Site, Pyungchon-Dong 896, Dongan-Gu
  - Novo Nordisk Investigational Site, Seongnam-si
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon
  - Novo Nordisk Investigational Site, Suwon-si, Gyeonggi-do
  - Novo Nordisk Investigational Site, Ulsan
  - Novo Nordisk Investigational Site, Wŏnju

REFERENCES:
- [Derived] Lee BW, Ahn KJ, Cho HC, Lee EY, Min K, Dahaoui A, Jeong JS, Lim HJ, Jang HC. Safety and Clinical Outcomes of Insulin Degludec in Korean Patients with Diabetes in Real-World Practices: A Prospective, Observational Study. Diabetes Ther. 2023 Oct;14(10):1659-1672. doi: 10.1007/s13300-023-01448-8. Epub 2023 Jul 19. PMID 37468685
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com